CLINICAL TRIAL: NCT02386059
Title: A Multicenter Randomized Trial to Evaluate the Efficacy and Safety of Three Different Prophylactic Treatments of Postoperative Nausea and Vomiting in Patients Undergoing Vitrectomy Under Local Anesthesia
Brief Title: Prevention of Postoperative Nausea and Vomiting in Patients Undergoing Vitrectomy Under Local Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, REIBALDI MICHELE, Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UCatania
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: ondansetron; dexamethasone; vitrectomy; local anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PLACEBO Group (Placebo Comparator): Received normal saline
  Interventions: Drug: PLACEBO
- DEXAMETHASONE Group (Active Comparator): Received 4 mg Dexamethasone.
  Interventions: Drug: Dexamethasone
- ONDANSETRON (Active Comparator): Received 4 mg Ondansetron
  Interventions: Drug: Ondansetron
- DEXAMETHASONE + ONDANSETRON (Active Comparator): Received 4mg Dexamethasone + 4mg Ondansetron
  Interventions: Drug: Dexamethasone + Ondansetron

INTERVENTIONS:
Drug: PLACEBO — received normal saline, intravenously
  Arms: PLACEBO Group
Drug: Dexamethasone — 4 mg, intravenously, at the start of surgery
  Arms: DEXAMETHASONE Group
Drug: Ondansetron — 4 mg, intravenously, 15 minutes before the end of surgery.
  Arms: ONDANSETRON
Drug: Dexamethasone + Ondansetron — 4 mg dexamethasone, intravenously at the start of surgery and 4 mg ondansetron intravenously 15 minutes before the end of surgery.
  Arms: DEXAMETHASONE + ONDANSETRON

SUMMARY:
Vitreoretinal surgery is associated with a considerable incidence of postoperative nausea and vomiting (PONV), which is reported to be as high as 60%. Reasons for this high incidence may be the long duration of surgery and anesthesia and the high degree of manipulation of the eye. Postoperative vomiting after vitrectomy is an important risk factor for the onset of several complications, such as suprachoroidal hemorrhage, with disastrous visual consequences.

To date there is no evidence as to the possible protective effect of anti-emetic therapy with regard to interventions of vitrectomy performed under local anesthesia.

In this prospective, randomized, multicenter, double blind study, we evaluated the efficacy of Ondansetron alone, Dexamethasone alone and in combination in controlling nausea and vomiting in patients undergoing vitrectomy under local anesthesia.

DETAILED DESCRIPTION:
Patients were randomly stratified to receive 1 of 4 prophylactic antiemetic treatments (3 pharmaceutical treatment and 1 placebo) in a double-blind manner at the start of the surgery and 15 minutes before the end of surgery.

The syringes were prepared by a third, neutral person not involved in the perioperative care of the patient, immediately before the start of anesthesia.

All vitrectomy surgeries were performed, in each unit,under local anesthesia by a retrobulbar block.

Each patients was observed and treated during a period of 24 hours after the surgery. For patients who have nausea and vomiting despite the antiemetic prophylaxis, will be given a rescue dose of 4 mg ondansetron IV.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older with an American Society of Anesthesiologists (ASA) physical status of I to II
* Scheduled for vitrectomy under local anesthesia

Exclusion Criteria:

* Hypersensitivity to study drug or rescue medication
* Preoperative score for nausea greater than 4 out of 10 points
* Subjects who suffer from chronic nausea and/or vomiting
* Severe hepatic insufficiency (Child-Pugh score > 9)
* Other antiemetic within 12 hours prior to surgery
* Patients unable to undergo a local anesthetic
* Subjects with clinically significant or unstable cardiac, respiratory, hepatic, renal, or other major organ system disease
* Psychotic illness or depression
* Addiction to illicit substances or alcohol
* Non-psychotic emotional disorders
* Pregnant or lactating
* Subjects who, in the opinion of the investigator, would experience an unacceptable risk from administration of study drug

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
• Proportion of patients with Complete Response (no nausea, no vomiting, no retching, and no use of rescue medication) during the first 24 hours after surgery | 1-24 hours post-operatively

SECONDARY OUTCOMES:
• Standardized score of nausea and/or vomiting severity if PONV occurs. | 1-24 hours post-operatively
• Pain score during the immediate post-operative period. | 1-24 hours post-operatively
• Number of antiemetic rescue medications given postoperatively. | 1-24 hours post-operatively
• Rates of known side effects. | 1-24 hours post-operatively

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Federico II University, Naples, Italy
  - University of Sassari, Sassari, Sardinia
  - University of Catania, Catania, Sicily
  - Polytechnic University of Marche, Ancona, The Marches